CLINICAL TRIAL: NCT01346618
Title: A Comparison of Bone Age Assessment by an Ultrasound Apparatus (SonicBone) and the X-ray Based Grulich and Pyle Method
Brief Title: The Validity of Bone Age Assessment by an Ultrasound Apparatus (SonicBone)
Status: Completed | Type: Observational
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Marianna Rachmiel, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 11/11
Record Dates: First submitted 2011-04-25; First posted 2011-05-03 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Bone Age
Keywords: bone age; children; x-ray; ultrasound; ultrasound based method; safe; valid; reproducable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children ages 4-17 years: Participants are children and youth ages 4-17 years (inclusive) who performed or will perform a X-ray of the left hand for bone age assessment as part of any clinical work up, within 2 months of enrollment in this study.

SUMMARY:
Bone age assessment is currently an important tool in final height implication in children. It is an important tool in the phases of investigation and treatment of short stature, tall stature, pubertal timing and various endocrinological pediatric situations. It is currently assessed using hand x-ray. This method has several limitations, including: requirement of specialized medical staff to interpret results, exposure radiation and usage of equipment which is only in radiology centers. The investigators aim to study a new equipment, radiation free, with simple and swift operation which provides an immediate answer, no need for an experienced observer, a mobile equipment with easy accessibility. The aim of the study is to assess its reproducibility, validity and safety compared to the x-ray method.

The investigators hypothesize it is as accurate and valid.

DETAILED DESCRIPTION:
Skeletal maturity assessment, defined also as bone age (BA), has an important role in pediatrics and pediatric endocrinology, used mainly for evaluating growth and puberty related endocrine disorders. Repeated BA assessment is important during the follow up of children with short stature, with precocious puberty and those treated by growth promoting medications.

The most commonly used method used for determining skeletal maturity, and thus BA is based on comparison of a hand and wrist radiographs to a standard series of representative films in the "Radiographic atlas of skeletal development of the hand and wrist" by Greulich and Pyle (GP), which has been issued several decades ago. Among the disadvantages and drawbacks in this BA assessment method are: the obligatory need for using radiology units that are often available only in special facilities or hospitals, not available at the physicians office, the exposure to ionizing radiation, and the known limitation of the method for the need of an endocrinologist to assess the BA, with a known large inter observers variability of the BA interpretation.

The suggested method in this study is based on ultrasound technology, and therefore it is quick, objective, and radiation-free. It delivers an immediate non biased result without the need to rely on an observer's evaluation of the hand radiograph and without the need for a specialized radiology facility.

This technique was innovated in order to find an efficient, convenient and non radiation based method of skeletal maturity assessment for the primary care physician that can be performed in an office setting.

The aim of this study is to establish a correlation algorithm between the BA assessment by an ultrasound apparatus (SonicBone) and the X-ray based assessment using Grulich and Pyle method, and to evaluate the validity and reproducibility of the apparatus, The design of the study is to perform a concomitant skeletal maturation assessment by reading of a hand X-ray radiograph by 3 experienced observers using the GP method, and by the ultrasound technique using the SonicBone apparatus. Skeletal maturation assessment will be performed in females and males at various age groups.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-17 years old
* Children who performed or will perform a hand x-ray as part of their clinical work up within 2 months from study enrolment
* A signed Informed Consent Form that was obtained from at least one parent or legal guardian and an audio approval by the other (phone call), if available, prior to ultrasound study.
* An assent from the child to perform the SonicBone's BA device reading

Exclusion Criteria:

* Children taking any medication that might change bone metabolism or mineralization within the last year (glucocorticosteroids, sex steroids, oral contraceptives, anticonvulsants, calcium and vitamin D in superphysiological doses)
* Children with suspected bone diseases or multiple fractures.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are children and youth ages 4-17 years (inclusive) who performed or will perform a X-ray of the left hand for bone age assessment as part of any clinical work up, within 2 months of enrollment in this study.
  Participants will be recruited according to advertising the study amongst pediatricians, pediatric endocrinologists and from the pediatric population who visits the pediatric endocrine clinic, endocrine testing room, adolescent medicine clinic, or being hospitalized at the pediatric division, Assaf Haroffeh Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
BA assessment readings by the SonicBone's BA device compared to the traditional GP method based reading of left hand x-ray and their reproducibility | 9 months

SECONDARY OUTCOMES:
The number of participants experiencing adverse side affects | 9 months
  Symptoms of pain, local erythema, syncope or pruritis will be assessed. Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Rachmiel, MD, Principal Investigator — Assaf Haroffeh Medical Center
Locations (1):
- Assaf Haroffeh Medical Center, Ẕerifin, Israel